CLINICAL TRIAL: NCT02081144
Title: Texting to Promote Tobacco Abstinence in Emergency Department Smokers: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1401013302; R01CA141479 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Smoking; Tobacco Abstinence
Keywords: Standard Care Condition; Texting + NRT Condition
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Condition (No Intervention): Control or Standard Care condition. No intervention will be provided.
- Texting + NRT Condition (Experimental): Enrollment in NCI's Smokefree TXT Program 4 weeks of Nicotine Replacement Patches 4 weeks of Nicotine Replacement Gum Faxed Referral CT Smokers Quitline
  Interventions: Other: Smokefree TXT Program; Drug: nicotine replacement patches; Drug: Nicotine Replacement Gum; Behavioral: Faxed Referral CT Smokers Quitline

INTERVENTIONS:
Other: Smokefree TXT Program — The SmokeFreeTxt program is a library consisting of ~130 brief messages that can be proactively sent to smokers' cellphones using software developed and maintained by NCI. The message content is informed by principles of cognitive behavioral therapy. They are sent to smokers at random times of day (during normal waking hours), up to 5 messages per day.
  Arms: Texting + NRT Condition
Drug: nicotine replacement patches — Subject will be given 4 weeks of Nicotine Replacement Patches, based on the amount he/she is smoking at baseline.
  Arms: Texting + NRT Condition
Drug: Nicotine Replacement Gum — Subjects will be given 10 pieces of 2mg Nicotine Replacement Gum x 28 days.
  Arms: Texting + NRT Condition
Behavioral: Faxed Referral CT Smokers Quitline — A faxed referral will be sent to the CT Smokers Quitline for the subject.
  Arms: Texting + NRT Condition

SUMMARY:
This is a pilot study to test the feasibility of conducting a text based smoking cessation trial with Emergency Department patients who are smokers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have smoked >= 100 cigarettes lifetime
* describe themselves as every or some day smokers
* are able to give written informed consent
* reside in Connecticut
* own a cell phone with texting capability.

Exclusion Criteria:

* inability to read or understand English
* currently receiving formal tobacco dependence treatment
* current use of tobacco cessation products (patch, gum, inhaler, nasal spray, lozenge, e-cigarette)
* currently using Zyban (bupropion), Wellbutrin (bupropion) or Chantix (varenicline) for smoking cessation
* current suicide or homicide risk
* current psychotic disorder
* life-threatening or unstable medical or psychiatric condition
* does not have phone with CT area code and with texting capability
* lacks capacity to give informed consent
* leaving the ED against medical advice
* pregnant, nursing, or trying to conceive
* incarcerated
* resides in an extended care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Survey of satisfaction and usage of Smokefree TXT Program | 1 month post enrollment
  Study team will develop a survey to assess both subjects' satisfaction with the Smokefree TXT Program and ease of use.

SECONDARY OUTCOMES:
7 day point prevalence abstinence | 1 month post enrollment
  7 day point prevalence abstinence will be assessed by asking if the subject has smoked even a puff in the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Bernstein, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States